CLINICAL TRIAL: NCT04823793
Title: A Fecal DNA Methylation Test for Colorectal Cancer Screening Using Multitarget Real-Time PCR Method-A Observational, Prospective Study
Brief Title: Fecal DNA Methylation Test for Colorectal Cancer Screening
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Yi-Chiao Cheng, Attending surgeon, division of colon and rectal surgery, Tri-Service General Hospital
Other Study IDs: A202105054
Record Dates: First submitted 2021-03-15; First posted 2021-04-01 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Colorectal Cancer; Colorectal Adenoma
Keywords: Fecal immunochemical testing; Methylation; Stool; Colonoscopy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — At least 40 specimens from participants with healthy colon at least 40 specimens from participants with adenoma/colorectal cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy group : Stool specimens from participants with healthy colon: Stool specimens will be collected from participants before having a colonoscopy.
  If the participant's colon has a healthy colon without any cancerous lesion, the stool specimen will be included in the healthy group.
  Interventions: Diagnostic Test: Stool DNA methylation detection
- Disease group : Stool specimens from participants with adenoma/colorectal cancer: Stool specimens will be collected from participants before having a colonoscopy.
  If the participant's colon has precancerous lesion, such as adenoma, the stool specimen will be included in the disease group.
  Also, specimens from confirmed colorectal cancer patients are included in the disease group.
  Interventions: Diagnostic Test: Stool DNA methylation detection

INTERVENTIONS:
Diagnostic Test: Stool DNA methylation detection — Stool specimens are collected from participants in the outpatient department or the inpatient department. Both FIT and stool DNA real-time PCR are performed simultaneously. To improve the sensitivity and specificity of the colorectal cancer screening, this study enrolls multiple candidate genes to distinguish whether the participant has a high risk of colorectal cancer.

SUMMARY:
This is an observational, prospective study using fecal DNA methylation test to define the risk of suffering from advanced adenoma or colorectal cancer (CRC) compared to colonoscopy and fecal immunochemical test (FIT).

This study recruits at least 80 participants, including 40 people of healthy controls, 20 people with adenoma, and 20 people with CRC, which were confirmed by colonoscopy. All fecal specimens from participants will be examined by FIT and multi-methylated target gene detection through real-time quantitative methylation-specific PCR (qMSP).

The objective of this study is to evaluate the sensitivity and specificity of multi-methylated target PCR compared with the FIT and confirm the examination results through colonoscopy.

DETAILED DESCRIPTION:
The incidence rate and the mortality rate of colorectal cancer (CRC) have been steadily increasing worldwide. Early detection of CRC can provide great opportunities to help patients, increasing their 5-year survival rate. Colonoscopy has been considered as the golden standard of CRC screening method, but the invasive procedures cannot be widely adapted by recipients.

Nowadays, the most common CRC screening method is fecal immunochemical test (FIT) which is a cost-effective and non-invasive approach. The sensitivity of FIT for CRC detection is about 80%, but only 20% for adenoma.

The methylation level of candidate genes are determined by qMSP to estimate the risk of colorectal cancer. This study implements fecal DNA methylation test and fecal immunochemical test simultaneously to evaluate whether the fecal DNA methylation test can improve the detection rate of adenoma and CRC.

ELIGIBILITY:
Inclusion Criteria:

* Participants with age over 40 but under 80, who need to take colonoscopy or diagnostic confirmed colorectal cancer patient.

Exclusion Criteria:

* Participants who are undergoing cancer treatments or have diagnosed with cancer, received cancer treatment in the past.
* Participants who have received any cancer treatments, including chemotherapy and radiotherapy before taking surgery.
* Participants have received any surgery for colorectal cancer in the past.
* Pregnant women or nursing women.

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy group :
  Participants without any cancerous lesion in their colon
  Disease group :
  Participants with adenoma or colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-03-31 (Actual); Primary Completion 2023-03-20 (Estimated); Study Completion 2023-03-20 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of methylation biomarker and FIT for adenoma and colorectal cancer screening | 6 months
  In this study, we estimate the sensitivity and specificity of methylation biomarker isolated from participant's stool DNA and perform FIT simultaneously.
  The Ct values of candidate genes and GAPDH (reference gene) are determined by real-time PCR. The delta Ct values are calculated by Ct value of candidate gene - Ct value of GAPDH. Furthermore, the cut-off value of each candidate gene was determined based on the Receiver Operating Characteristic curve.
  If the value of Fecal immunochemical test is more than 100 ng Hb/ml, the stool is considered as positive with fecal occult blood.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Chiao Cheng, MD, Principal Investigator — Tri-Service General Hospital
Locations (1):
- Tri-Service General Hospital, National Defense Medical Center, Taipei, Taiwan